CLINICAL TRIAL: NCT06008210
Title: Effects of a Decision Support Intervention on End-of-life Care Planning in Patients With Advanced Chronic Obstructive Pulmonary Disease and Their Family Members: A Mixed Method Approach
Brief Title: A Decision Aid on End-of-life Care for Patients With Advanced COPD and Their Family
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Health Bureau, Hong Kong (Other Government)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Helen YL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14118622
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe
Keywords: Advance Care Planning; Decision making; End-of-life care

STUDY DESIGN:
Intervention Model Description: A parallel two-arm single-blinded randomised controlled trial will be conducted.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Decision Support Intervention
  Interventions: Behavioral: Decision Support Intervention
- Control Group (Active Comparator): Health coaching
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Decision Support Intervention — The participants will receive two 60-minute consultation sessions delivered by a trained nurse in four weeks at home. Participant's family members will be encouraged to attend the sessions. In the first session, the nurse will explore the participant's understanding of the current health condition, introduce the concept of advance care planning and discuss their decisional needs for end-of-life care decision-making. In the second session, the nurse will ask the participants to complete a value clarification exercise individually.
  Arms: Intervention Group
Behavioral: Health Coaching — The participants will receive two 60-minute health coaching sessions delivered by a trained nurse in four weeks at home. This intervention will focus on lifestyle modification and self-care management unrelated to the tested intervention content or outcomes.
  Arms: Control Group

SUMMARY:
This study aims to support EOL decision-making in patients with advanced COPD and their family members. A parallel two-arm single-blinded randomised controlled trial will be conducted to evaluate the effects of a specific decision support intervention. A total of 226 patients with advanced COPD and their designated family members will be recruited from hospital wards and outpatient clinics.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive life-limiting condition. However, patients with advanced COPD and their family members generally are unprepared for end-of-life (EOL) situations. The Ottawa Decision Support Framework model is adopted to address the patients' decisional needs for the difficult decisions in EOL care. The participants will be randomly allocated to either the intervention group to receive the decision support intervention or the control group to receive general health coaching. Outcomes will be measured at baseline and 1- and 6-month post-allocation. Subsequently, a descriptive qualitative study will be conducted with a subsample of 30 dyads to explore how the intervention influenced the study outcomes.

ELIGIBILITY:
Inclusion Criteria of patients:

* are aged 50 years or over
* have been diagnosed with COPD
* are cognitively sound (scored > 5 on the validated Abbreviated Mental Test (Hong Kong version) [AMT-HK])
* meet at least two of the six specific clinical indicators related to advanced COPD in the Gold Standards Framework (GSF) Proactive Identification Guidance, 6th Edition
* can nominate a family member who would take part in their healthcare decision- making.

Inclusion Criteria of patients' family members:

* are aged 18 years or over,
* can communicate in Cantonese,
* have at least one personal contact per week with the patient in the past 6 months and
* are willing to join the study. Family members will be excluded if they score < 6 on the AMT-HK or are expecting to leave Hong Kong within the next 6 months.

Exclusion Criteria:

* non-communicable due to a severe hearing impairment, dysphasia or a language barrier;
* are receiving palliative care services or
* have already completed ACP or an advance directive.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict at T0 | Baseline
  Decisional conflict regarding EOL care measured using The SURE test. It includes four items to be rated on a dichotomous format, with 0 (no) or 1 (yes). The total score ranged from 0 to 4, with a higher score means less decisional conflict.
Decisional conflict at T1 | 1-month post allocation
  Decisional conflict regarding EOL care measured using The SURE test. It includes four items to be rated on a dichotomous format, with 0 (no) or 1 (yes). The total score ranged from 0 to 4, with a higher score means less decisional conflict.
Decisional conflict at T2 | 6-month post allocation
  Decisional conflict regarding EOL care measured using The SURE test. It includes four items to be rated on a dichotomous format, with 0 (no) or 1 (yes). The total score ranged from 0 to 4, with a higher score means less decisional conflict.

SECONDARY OUTCOMES:
Self-efficacy for ACP at T0 | Baseline
  Self-efficacy for ACP measured using the 3-item Self-efficacy subscale of the ACP Engagement Survey. Participants will rate their level of self-efficacy regarding three ACP actions - namely, appointing a surrogate and discussing EOL care with a surrogate and with medical doctors - using a five-point Likert scale. A higher score indicates a higher level of self-efficacy.
Self-efficacy for ACP at T1 | 1-month post allocation
  Self-efficacy for ACP measured using the 3-item Self-efficacy subscale of the ACP Engagement Survey. Participants will rate their level of self-efficacy regarding three ACP actions - namely, appointing a surrogate and discussing EOL care with a surrogate and with medical doctors - using a five-point Likert scale. A higher score indicates a higher level of self-efficacy.
Self-efficacy for ACP at T2 | 6-month post allocation
  Self-efficacy for ACP measured using the 3-item Self-efficacy subscale of the ACP Engagement Survey. Participants will rate their level of self-efficacy regarding three ACP actions - namely, appointing a surrogate and discussing EOL care with a surrogate and with medical doctors - using a five-point Likert scale. A higher score indicates a higher level of self-efficacy.
Readiness for ACP at T0 | Baseline
  Readiness for completing the aforementioned three ACP actions based on the ACP Engagement Survey. Participants will rate their readiness using a five-point scale, from 1 (never thought about it) to 5 (completed already). The total score ranged from 4 to 20. A higher score indicates a higher level of readiness.
Readiness for ACP at T1 | 1-month post allocation
  Readiness for completing the aforementioned three ACP actions based on the ACP Engagement Survey. Participants will rate their readiness using a five-point scale, from 1 (never thought about it) to 5 (completed already). The total score ranged from 4 to 20. A higher score indicates a higher level of readiness.
Readiness for ACP at T2 | 6-month post allocation
  Readiness for completing the aforementioned three ACP actions based on the ACP Engagement Survey. Participants will rate their readiness using a five-point scale, from 1 (never thought about it) to 5 (completed already). The total score ranged from 4 to 20. A higher score indicates a higher level of readiness.
Family members' engagement in ACP at T0 | Baseline
  Family members' engagement in ACP will be measured by using the 17-item ACP Engagement Survey for Surrogate Decision Makers. Participants will rate their level of engagement using a five-point scale, from 1 (least) to 5 (highest). The total score ranged from 17 to 85. A higher score indicates a higher level of engagement.
Family members' engagement in ACP at T1 | 1-month post allocation
  Family members' engagement in ACP will be measured by using the 17-item ACP Engagement Survey for Surrogate Decision Makers. Participants will rate their level of engagement using a five-point scale, from 1 (least) to 5 (highest). The total score ranged from 17 to 85. A higher score indicates a higher level of engagement.
Family members' engagement in ACP at T2 | 6-month post allocation
  Family members' engagement in ACP will be measured by using the 17-item ACP Engagement Survey for Surrogate Decision Makers. Participants will rate their level of engagement using a five-point scale, from 1 (least) to 5 (highest). The total score ranged from 17 to 85. A higher score indicates a higher level of engagement.
End-of-life care preferences at T1 | 1-month post allocation
  End-of-life care preferences will be determined using the adapted Life-Support Preferences Questionnaire. Participants will be asked to indicate whether they would accept cardiopulmonary resuscitation, mechanical ventilator and tube feeding if they become seriously ill and mentally incapacitated. There are three options: yes, no and uncertain. In addition, they will be asked to indicate their preferred goal of end-of-life care. The available options are maintain life at all costs, maintain comfort and uncertain. There is no scoring for the responses.
End-of-life care preferences at T2 | 6-month post allocation
  End-of-life care preferences will be determined using the adapted Life-Support Preferences Questionnaire. Participants will be asked to indicate whether they would accept cardiopulmonary resuscitation, mechanical ventilator and tube feeding if they become seriously ill and mentally incapacitated. There are three options: yes, no and uncertain. In addition, they will be asked to indicate their preferred goal of end-of-life care. The available options are maintain life at all costs, maintain comfort and uncertain. There is no scoring for the responses.
Advance directives at T2 | 6-month post allocation
  Participants will be asked if they have completed advance directives in the past six months.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Chan, Ph.D., Principal Investigator — Chinese University of Hong Kong
Locations (2):
- China (2):
  - Prince of Wales Hospital, Hong Kong
  - Tai Po Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request